CLINICAL TRIAL: NCT00442273
Title: Comparison of Autologous Serum and Umbilical Cord Serum Eyedrops for Dry Eye Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCS-0001
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

INTERVENTIONS:
Drug: Umbilical cord serum eyedrops
Drug: Autologous serum eyedrops

SUMMARY:
To compare the therapeutic effect between autologous serum and umbilical cord serum eyedrops in the treatment of severe dry eye syndrome.

DETAILED DESCRIPTION:
Ninety-two eyes of 48 patients with severe dry eye syndrome (34 eyes of 17 patients with Sjögren's syndrome and 58 eyes of 31 patients with non-Sjögren's syndrome) were treated with either 20% autologous serum (41 eyes of 21 patients) or umbilical cord serum eyedrops (51 eyes of 27 patients). Symptom scoring, corneal sensitivity test, tear film break-up time (BUT), Schirmer test, tear clearance rate (TCR), corneal fluorescein staining, and conjunctival impression cytology were performed before and 1 month and 2 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe dry eye syndrome who were refractory to conventional treatments and had symptoms of dry eye for more than 3 months
* Low tear film break-up time (BUT, < 5 sec)
* Low Schirmer test (5 mm)
* Positive fluorescein or rose bengal vital staining (≥ 3)

Exclusion Criteria:

* Active ocular infection or inflammation not associated with dry eye
* Contact lens wear
* Ocular allergy
* Ocular surgery within the recent 3 months
* Lid or lash abnormalities
* Pregnant or lactating women

Ages: 20 Years to 61 Years | Sex: All
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kyung chul Yoon, M.D., Study Director — Chonnam natianl university hospital
Locations (1):
- Chonnam national university hospital, Gwangju, South Korea